CLINICAL TRIAL: NCT06781853
Title: Evaluating the Effectiveness of Cognitive Behavioral Therapy for Muscle Dysmorphia and Steroid Abuse: A Randomized Controlled Trial
Brief Title: CBT for Muscle Dysmorphia and Steroid Abuse: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Collaborators: Beykoz University (Other); Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Selami Varol Ülker, Assistant Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61351342/20-318
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Body Dysmorphic Disorder; Steroid Abuse; Body Dysmorphic Disorder (BDD), Subtype: Muscle Dysmorphia
Keywords: Cognitive Behavioral Therapy (CBT); Muscle Dysmorphia; Body Dysmorphic Disorder (BDD); Steroid Abuse; Performance-Enhancing Drugs (PEDs)
MeSH Terms: conditions — Body Dysmorphic Disorders; Brachydactyly, Type D | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study employs a randomized controlled trial (RCT) with a parallel assignment model to evaluate the effectiveness of cognitive behavioral therapy (CBT) for men diagnosed with muscle dysmorphia (MD) and steroid/PED abuse. Participants will be randomly assigned to an experimental group (12 weekly online CBT sessions) or a control group (no intervention). Assessments will occur at baseline, post-intervention, and three-month follow-up to measure changes in MD symptoms, psychological distress, and related behaviors. Therapists will be supervised by clinical psychologists and psychiatrists, with adherence monitored by an external committee to ensure fidelity to the CBT protocol. This design ensures a robust evaluation of the intervention's impact while addressing accessibility and stigma-related barriers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT Interventional Group (Experimental): Participants in this group will receive 12 weekly one-on-one cognitive behavioral therapy (CBT) sessions, each lasting 50 minutes, delivered online via Microsoft Teams. The intervention will target symptoms of muscle dysmorphia (MD), maladaptive thoughts, and behaviors related to steroid and performance-enhancing drug (PED) abuse. Therapy will be conducted by three assistant professors in psychology supervised by senior author psychiatrist.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control Group (No Intervention): Participants in this group will not receive any intervention during the study period. They will complete the same assessments as the experimental group at baseline, post-intervention, and three-month follow-up to evaluate changes in muscle dysmorphia symptoms, psychological distress, and related behaviors for comparison. After the study, participants in this group will be offered an intensive 8-session CBT program if requested.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The intervention consists of 12 weekly one-on-one online CBT sessions, each lasting 50 minutes, delivered via Microsoft Teams. The sessions will focus on addressing symptoms of muscle dysmorphia (MD), maladaptive thought patterns, and behaviors associated with steroid and performance-enhancing drug (PED) use. The therapy is based on structured CBT techniques and will include psychoeducation, cognitive restructuring, behavioral experiments, and relapse prevention strategies. The sessions will be conducted by trained clinical psychology master's students under the supervision of experienced clinical psychologists and a psychiatrist. The intervention is designed to reduce MD symptoms and improve psychological well-being.
  Arms: CBT Interventional Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of cognitive behavioral therapy (CBT) in treating muscle dysmorphia (MD) under body dysmorphic disorder (BDD) and steroid/performance-enhancing drug (PED) abuse in men aged 18-65 who regularly attend the gym. The main questions it aims to answer are:

Does CBT reduce the symptoms of muscle dysmorphia in this population? Does CBT improve psychological well-being and reduce reliance on steroids or PEDs? Researchers will compare participants receiving CBT to a control group that does not receive any intervention to determine the therapy's effectiveness.

Participants will:

Undergo a formal diagnosis of muscle dysmorphia (Under BDD) and steroid/PED abuse based on DSM-5-TR criteria through online clinical interviews.

Complete 12 weekly one-on-one online CBT sessions (50 minutes each) for those in the experimental group.

Complete psychological assessments at three time points: before the intervention, after the intervention, and at a 3-month follow-up.

This study uses validated scales to measure changes in symptoms of MD, psychological distress, and other related outcomes. The results will help determine if CBT is an effective treatment for muscle dysmorphia and associated steroid/PED abuse.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate the effectiveness of cognitive behavioral therapy (CBT) for men diagnosed with muscle dysmorphia (MD) under body dysmorphic disorder (BDD) and steroid or performance-enhancing drug (PED) abuse. Muscle dysmorphia is a subtype of BDD characterized by a pathological preoccupation with insufficient muscularity, often accompanied by steroid/PED use. Despite the physical and psychological risks associated with these behaviors, individuals with MD and steroid abuse rarely seek treatment due to stigma and the psychological effects of steroid use.

Study Design:

The trial will recruit male participants aged 18-65 who regularly attend the gym (at least three times per week) and have been using steroids or PEDs for at least one year. Recruitment will be conducted across 6 districts in Istanbul, targeting a diverse range of socioeconomic populations. Survey teams will approach gym-goers outside fitness clubs to introduce the study, explain its confidentiality, and emphasize the benefits of participation, including free psychiatric diagnosis and CBT sessions.

Participants will be asked to complete a sociodemographic questionnaire, and formal diagnoses of muscle dysmorphia and steroid/PED abuse will be made via online clinical interviews conducted by a psychiatrist using DSM-5-TR criteria.

Randomization and Intervention:

Participants who meet the inclusion criteria will be randomly assigned to one of two groups:

Experimental Group: Participants will receive 12 weekly one-on-one CBT sessions (50 minutes each) conducted online via Microsoft Teams. Therapy will be structured to address MD symptoms, maladaptive thought patterns, and behaviors associated with steroid/PED use.

Control Group: Participants will not receive any intervention during the study period.

Therapy sessions will be delivered by 3 side-principle investigators (authors of the study) and assistant professors in psychology who have BDD/MD and steroid abuse experinces . The therapy process will be supervised by psychiatry professor (one of the author) ensure adherence to the treatment protocol.

Outcome Measures:

Participants in both groups will be assessed at three time points: baseline (pre-intervention), post-intervention, and three-month follow-up. The following validated scales will be used:

Muscle Dysmorphic Disorder Inventory (MDDI) Patient Health Questionnaire (PHQ) Kessler Psychological Distress Scale (K10) Bodybuilder Image Grid (BIG) Eating Disorder Examination Questionnaire (EDE-Q) Exercise Addiction Inventory (EAI)

Monitoring and Supervision:

To maintain fidelity to the CBT protocol, an external monitoring committee will review recordings of therapy sessions. The committee will include two CBT-trained clinical psychologists, one clinical psychology PhD assistant professor, and one psychiatrist. Feedback will be provided to therapists to ensure consistency and adherence to the protocol.

Challenges and Mitigation:

Recognizing the stigma associated with steroid use and MD, the study incorporates strategies to build trust and encourage participation, including emphasizing confidentiality, offering free psychiatric diagnosis and therapy, and using trained survey teams to engage participants effectively. To minimize dropout rates, reminders and follow-ups will be implemented throughout the study period.

Significance:

This trial aims to address a critical gap in the treatment of muscle dysmorphia and steroid/PED abuse. By evaluating the efficacy of structured CBT delivered online, the study will provide valuable insights for developing accessible and effective interventions for this underserved and stigmatized population.

ELIGIBILITY:
Inclusion Criteria:

Male participants aged 18-65. Regular gym attendance (minimum three times per week). Use of steroids or performance-enhancing drugs (PEDs) for at least one year. Formal diagnosis of muscle dysmorphia (MD) under body dysmorphic disorder (BDD) and steroid/PED abuse, based on DSM-5-TR criteria.

Willingness to participate in 12 weekly one-on-one online cognitive behavioral therapy (CBT) sessions.

Ability to provide informed consent and complete assessments at baseline, post-intervention, and three-month follow-up.

Exclusion Criteria:

Diagnoses of substance use disorders (e.g., heroin, cannabis). Diagnoses of bipolar disorder or antisocial personality disorder. Use of steroids or PEDs for medical purposes. Use of medications that could interfere with the study outcomes. Participation in any other psychotherapy or psychological intervention during the study period.

Inability to access the internet or participate in online therapy sessions.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in Muscle Dysmorphia Symptoms | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks).
  Change in muscle dysmorphia symptoms, as measured by the Muscle Dysmorphic Disorder Inventory (MDDI), from baseline to post-intervention and three-month follow-up.

SECONDARY OUTCOMES:
Reduction in Psychological Distress | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks).
  Change in psychological distress, as measured by the Kessler Psychological Distress Scale (K10), from baseline to post-intervention and three-month follow-up.
Improvement in General Psychological Well-being | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks).
  Change in general psychological well-being, assessed using the Patient Health Questionnaire (PHQ), from baseline to post-intervention and three-month follow-up.
Reduction in Risky Body Image Behaviors | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks).
  Change in risky body image behaviors, as measured by the Bodybuilder Image Grid (BIG), from baseline to post-intervention and three-month follow-up.
Reduction in Eating Disorder Symptoms | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks).
  Change in eating disorder symptoms, as measured by the Eating Disorder Examination Questionnaire (EDE-Q), from baseline to post-intervention and three-month follow-up.
Reduction in Exercise Addiction Symptoms | Baseline, post-intervention (12 weeks), and three-month follow-up (24 weeks)
  Change in symptoms of exercise addiction, assessed using the Exercise Addiction Inventory (EAI), from baseline to post-intervention and three-month follow-up.

OTHER OUTCOMES:
Dropout Rates | End of the intervention phase (12 weeks).
  Percentage of participants in the experimental group who attend fewer than 75% of sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Selami Varol Ülker, Phd, Principal Investigator — Üsküdar University; Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi University; Eda Yılmazer, Phd, Principal Investigator — Beykoz University; Gokben Hızlı Sayar, Professor, Study Chair — Üsküdar University
Locations (1):
- Üsküdar University, İstanbul, Türkiye, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) related to the study's primary and secondary outcome measures will be shared with other researchers upon reasonable request. The shared data will include de-identified demographic information, baseline characteristics, and assessment scores. Data will be made available following publication of the study results and can be accessed by submitting a request to the corresponding author. Requests must include a detailed research proposal and comply with all applicable ethical and legal requirements. The data will be shared in a secure format to ensure participant confidentiality.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The IPD and supporting information will be available starting 6 months after publication of the study results and will remain accessible for 5 years.
Access Criteria: Access to the de-identified IPD and supporting information will be granted to qualified researchers upon reasonable request. Requests must include a detailed research proposal outlining the intended use of the data and compliance with applicable ethical and legal standards. Access will be provided after review and approval by the study's data-sharing committee. Researchers will be required to sign a data use agreement to ensure the confidentiality of the participants and appropriate use of the data. Requests can be submitted to the corresponding author via email.